CLINICAL TRIAL: NCT01069029
Title: Macular Hole and Cataract Extraction: Combined Surgery Versus Two Times Surgery
Brief Title: Combined Versus Successive Macular Hole and Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Pr Catherine Creuzot-Garcher, Ophthalmology Department CHU Dijon
Other Study IDs: Aurore 1
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2006-01

CONDITIONS: Macular Hole; Visual Acuity
Keywords: Macular Hole; Cataract surgery; Vitreoretinal surgery; Combined surgery; Idiopathic
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Combined surgery: Patient which underwent combined surgery of MH and cataract extraction
- Successive surgery: Patients which underwent the two successive procedures

SUMMARY:
The purpose of this study is to compare functional and anatomical results of a combined surgery and two time surgery for macular hole and cataract extraction in one hundred and twenty patients (120 eyes) with idiopathic Macular Hole (MH) and cataract in two academic centers.

DETAILED DESCRIPTION:
Main outcome measures were the assessment of visual acuity at 6 and 12 months,and the rate of closure of MH by OCT (optical coherence tomography).

ELIGIBILITY:
Inclusion Criteria:

* Macular Hole Stage 2,3,and 4
* Visual loss
* At least 18 years of age

Exclusion Criteria:

* Stage of Macular Hole Stage 1
* Macular hole post traumatism or associated with retinal detachment
* Diabetic retinopathy
* Glaucoma
* Age-related macular degeneration
* Myopia > 6 diopters
* Preoperative pseudophakia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic visual loss and needed vitrectomy for Macular Hole treatment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Post surgical procedure assessment of Visual acuity | 6 and 12 months post surgery

SECONDARY OUTCOMES:
Rate of closure of macular hole by OCT | at 6 and 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Creuzot-Gracher, MD, PhD, Principal Investigator — Ophthalmology unit CHU Dijon
Locations (1):
- Ophthalmology Unit CHU Dijon, Dijon, Burgundy, France

REFERENCES:
- [Derived] Muselier A, Dugas B, Burelle X, Passemard M, Hubert I, Mathieu B, Berrod JP, Bron AM, Creuzot-Garcher C. Macular hole surgery and cataract extraction: combined vs consecutive surgery. Am J Ophthalmol. 2010 Sep;150(3):387-91. doi: 10.1016/j.ajo.2010.04.008. Epub 2010 Jul 7. PMID 20615492